CLINICAL TRIAL: NCT01636310
Title: Multiple Cigarette Induced Changes in Hormone Function, Mood States and Behavior
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical studies stopped, pending funding
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Nancy Kishlar Mello, Director, Alcohol and Drug Abuse Research Center & Professor of Psychology (Neuroscience), Harvard Medical School, Mclean Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2005-p-002454
Record Dates: First submitted 2012-06-21; First posted 2012-07-10 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Female Smokers (Mid-Luteal Phase; cycle days 18-22) (Active Comparator)
  Interventions: Other: Nicotine
- Female Smokers (Early Follicular Phase; cycle days 4-8) (Active Comparator)
  Interventions: Other: Nicotine

INTERVENTIONS:
Other: Nicotine — Two doses of nicotine will be utilized: a commercially available, high-yield nicotine cigarette (Marlboro Red; Phillip Morris brand) and a denicotinized cigarette (Murty Pharmaceuticals Inc., Lexington, KY). The high dose cigarettes contain 15.48 mg of nicotine and 16 mg of tar based on analysis by the Massachusetts Department of Public Health (MDPH, 1998). The low nicotine cigarettes contain 1.1 mg of nicotine and deliver 0.1 mg of nicotine and 2.8 mg of tar based on analyses provided by the manufacturer.

SUMMARY:
The proposed clinical studies will analyze the interactions between nicotine, alterations in endocrine hormones, mood and cardiovascular measures. They also intend to examine the contribution of gender and menstrual cycle phase. These studies hypothesize that this novel focus on nicotine's rapid hormonal, cardiovascular and subjective effects will be important for developing novel biologic approaches to treatment for nicotine abuse and dependence as well as advancing our understanding of the neurobiology of nicotine reinforcement.

DETAILED DESCRIPTION:
Clinical studies are proposed to measure the covariance between nicotine-induced changes in endocrine, subjective and cardiovascular effects and the temporal concordance with increases in serum nicotine and cotinine levels. Possible gender and menstrual cycle phase influences on the effects of nicotine on HPA and HPG hormones have not been clearly delineated. Accordingly, we propose to compare the acute effects of nicotine in men and women, and to study women at the follicular and the luteal phases of the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 40 who currently smoke at least 15 cigarettes every day, and who fulfill DSM-IV diagnostic criteria for nicotine dependence (305.10) will be eligible for participation.
* No evidence of clinically significant disease based upon complete medical history and physical examination by a qualified physician.
* Absence of DSM-IV Axis I Disorders other than nicotine dependence (305.10) as measured by the Structured Clinical Interview (SCID).
* Routine laboratory blood tests including complete blood count, electrolytes, BUN and creatinine, liver function test, hepatitis panel and urinalysis will be performed. Laboratory parameters must be within the normal range. HBsAg must be negative but study participants who have hepatitis serology consistent with previous exposure to Hepatitis A, Hepatitis B, or Hepatitis C, but who do not have clinical and biochemical evidence of acute infection, will be acceptable.
* Hematocrit levels ≥ 35%.
* Serum pregnancy test (hCG beta subunit) results must be negative within 24 hrs of the study day.
* Normal ECG.
* A mean Body Mass Index (ratio of weight (W) to height (H) squared; W/H2=kg/m2) will be calculated. Women with a mean Body Mass Index (BMI) between 18.0-27.0 will be accepted.
* Study participants must be able to read, understand instructions and provide a valid informed consent.

Exclusion Criteria:

* Women with any lifetime DSM-IV Axis I disorder other than nicotine dependence will be excluded.
* Women who are pregnant as determined by laboratory testing for serum beta hCG will be excluded.
* Women who use hormonal contraceptive medications will not be accepted for participation because this would confound the hormonal measures.
* Women with clinically significant medical disorders will be excluded.
* A mean Body Mass Index (ratio of weight (W) to height (H) squared; W/H2=kg/m2) will be calculated. Women with a mean Body Mass Index (BMI) outside of the range of 18.0-27.0 will be excluded.
* Treatment seeking study participants will not be selected but will be referred to local smoking cessation programs.
* Women taking any OTC medications on a regular basis (with the exception of multivitamin formulas) or prescription medications will be excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2005-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Effects of Nicotine on the hypothalamic-pituitary-adrenal (HPA) axis | From baseline to study completion (approximatley 8 months for females)
  The investigators are examining the effects of smoked nicotine on serum nicotine levels and serum/plasma hormone levels.
Effects of Nicotine on the hypothalamic-pituitary-gonadal (HPG) axis | From baseline to study completion (approximately 8 months for females)
  The investigators are examining the effects of smoked nicotine on serum level nicotine and serum/plasma hormone levels.

SECONDARY OUTCOMES:
Effects of Nicotine on Mood States on the Visual Analog Scale | From baseline to study completion (approximately 8 months for females)
  The investigators are examining the effects of smoked nicotine on subjective states ("high," "like," "rush," "dizzy," etc.) as measured by a visual analog scale.
Effects of Nicotine on cardiovascular measures | From baseline to study completion (approximately 8 months for females)
  The investigators are examining the effects of smoked nicotine on cardiovascular measures, as measured by heart rate and blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Mello, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- Alcohol and Drug Abuse Research Center at McLean Hospital, Belmont, Massachusetts, United States